CLINICAL TRIAL: NCT04383652
Title: Collection of Coronavirus COVID-19 Outbreak Samples in New South Wales
Acronym: COSiN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: VISP2005
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult cohort: 1. Diagnosed with SARS-CoV-2 infection (COVID-19; by a registered diagnostic facility)
  2. Age 16 years or older
  3. Have provided informed consent
  Blood samples and clinical data related to COVID19 diagnosis, symptoms, and outcomes will be collected.
  Interventions: Other: Biological sample and clinical data collection
- Paediatric cohort: 1. Diagnosed with SARS-CoV-2 infection (COVID-19; by a registered diagnostic facility)
  2. Age less than 16 years
  3. Parent or caregiver has provided informed consent Blood samples and clinical data related to COVID19 diagnosis, symptoms, and outcomes will be collected.
  Interventions: Other: Biological sample and clinical data collection

INTERVENTIONS:
Other: Biological sample and clinical data collection — Plasma and serum will be collected at day 0, day 7, day 14, 1 month and 4 months post diagnosis. Clinical data related to COVID-19 diagnosis, symptoms, and outcomes will be collected.

SUMMARY:
The objectives of this study are to characterise immune responses in people with CoV-SARS-2 infection and use this knowledge to advance vaccine design, treatment options, and diagnostic reagents. Eligible participants will include people diagnosed with SARS-CoV-2 infection, and may include recently returned travellers and non-travellers in the community presenting to tertiary hospital healthcare facilities. Recruitment will be opportunistic, and sampling intensity may vary depending on the phase of the outbreak. Participants can be enrolled at any timepoint (up to 6 months) following diagnosis of SARS-CoV-2 infection (COVID-19). Blood samples and clinical data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Main cohort

  1. Diagnosed with CoV-SARS-2 infection
  2. 16 years of age or older
  3. Have provided informed consent Paediatric cohort

  <!-- -->

  1. Diagnosed with CoV-SARS-2 infection
  2. Less than 16 years of age
  3. Informed consent provided by parent or caregiver

     Exclusion Criteria:

     Main cohort

  <!-- -->

  1. 15 years of age or younger
  2. Inability or unwillingness to provide informed consent or abide by the requirements of the study Paediatric cohort

  <!-- -->

  1. 16 years of age or older
  2. Inability or unwillingness of parent or caregiver to provide informed consent or abide by the requirements of the study -

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be adults, adolescents or children diagnosed with COVID-19 and attending a major teaching hospital located in Sydney, New South Wales Australia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Coronavirus sequencing | 4 months post COVID-19 diagnosis.
  The viruses will be sequenced to to help understand epitope specificity

SECONDARY OUTCOMES:
Coronavirus culturing | 4 months post COVID-19 diagnosis.
  The viruses will then be either cultured to study the immune response against them in culture.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Martinello, Principal Investigator — Kirby Institute, UNSW Sydney; Rowena Bull, Principal Investigator — School of Medical Sciences, UNSW Sydney
Locations (9):
- Australia (9):
  - NSW Health Pathology, Randwick, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - Blacktown Hospital, Blacktown
  - Royal Prince Alfred Hospital, Camperdown
  - St Vincent's Hospital, Darlinghurst
  - Northern Beaches Hospital, Frenchs Forest
  - Royal North Shore Hospital, Saint Leonards
  - Westmead Hospital, Westmead

IPD SHARING:
Plan to Share IPD: No
Access to samples and data is governed by the Protocol Steering Committee. Requests can be made to the Committee (via the Principal Investigators).